CLINICAL TRIAL: NCT07051005
Title: A Feasibility Randomised Controlled Trial of Online Self-compassion Training Tailored for Adults Living With Type 1 and Type 2 Diabetes Mellitus
Brief Title: Feasibility of a Tailored Online Self-compassion Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Collaborators: Barts & The London NHS Trust (Other); Betsi Cadwaladr University Health Board (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ETH2425-0223
Record Dates: First submitted 2025-06-03; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus (T2DM)
Keywords: Diabetes; Online intervention; Compassion; Feasibility RCT
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All the outcome measures will be self-report questionnaires that will be completed by an online automated system with no involvement of the research team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Intervention (Experimental): Four Week Online Self-Compassion Course
  Interventions: Behavioral: Feasibility RCT of a tailored online self-compassion intervention
- Waitlist Control (No Intervention): Control participants will receive no intervention during the study but will be given the option of accessing the online self-compassion intervention after the study is complete.

INTERVENTIONS:
Behavioral: Feasibility RCT of a tailored online self-compassion intervention — This is a four-week online self-compassion course supplied by Balanced Minds. The researches of this study and an Expert by Experience have consulted with the owner of Balanced Minds to tailor this programme to people with diabetes.
  The self-help, self-compassion course is based on Compassionate Mind Training. This provides participants with opportunities to develop skills and attributes of compassion through a weekly 30-minute video on a specified topic, a 10-minute compassionate exercise that participants are encouraged to engage in daily for the week and a brief summary of the compassionate topic. The topics of the course are:
  The Foundations of Self-Compassion Developing your Compassionate Self Deepening the Compassionate Relationship with Yourself Self-compassion in Everyday Life.
  Arms: Online Intervention

SUMMARY:
The goal of this clinical trial is to examine the feasibility and acceptability of an online programme that is based on Compassionate Mind Training (CMT) over four-weeks. The programme intends to share information and strategies to reduce diabetes distress, self-criticism, and shame, and improve physical health in people who have Type 1 and Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
This pilot randomised controlled trial seeks to examine the feasibility and acceptability of online compassion training tailored for adults living with Type 1 and Type 2 diabetes. Participants will be randomised to either the compassion training course or a waitlist control group, in which participants will be offered the intervention at the end of the study. Four self-report measures will be administered online at baseline (weeks 0-1) and post-intervention (weeks 9-10). The indices of feasibility and acceptability that will be examined include: 1. ease of recruitment; 2. participant retention in the intervention; 3. participant retention in the study; 4. acceptability of the intervention; 5. outcome measure completion; 6. whether there is a preliminary signal of efficacy on the primary outcome measure (diabetes distress). These indices will be compared to progression criteria which determine whether the intervention is sufficiently feasible and acceptable to progress to a full-scale RCT in future research.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older.
* Diagnosed with Type 1 or Type 2 diabetes by a clinician in the NHS more than one year ago.
* Self-managing theircondition.
* Identified by their NHS team as needing support with their mental health due to diabetes-related distress.

Exclusion Criteria:

* <18
* Individuals experiencing a current mental health crisis, including severe depression, active suicidal thoughts, or acute psychosis
* Unable to read/speak English
* Gestational diabetes, Wolfram, and other rarer conditions
* Individuals currently experiencing severe substance abuse issues that could interfere with participation in the programme
* Individuals without reliable access to the internet and a compatible device (computer or smartphone).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited | 6 months following the start of recruitment
  The number of participants recruited over 6-months will be compared against the following progression criterion to assess the feasibility of recruitment: Green: 40-50; Amber 24-39; Red: <24.
Proportion of intervention group participants who complete at least half of the compassion training course intervention sessions | Weeks 2 to 8
  The proportion of participants who completed at least half of the intervention sessions will be compared against the following progression criterion to assess retention in the intervention: Green: ≥50%; Amber 25-49%; Red: <25%.
Proportion of study participants who remain in the study | Weeks 0 to 10
  The proportion of study participants who remain in the study will be compared against the following progression criterion to assess retention in the study: Green: ≥50%; Amber 25-49%; Red: <25%.
Compassion training course acceptability | Weeks 9 to 10
  Response to Likert type questions and content analysis of qualitative data will be compared against the following progression criterion to assess retention in the study: Green: the majority of intervention participants report the intervention is acceptable as it is or with minor adjustments; Amber: there are inconsistent reports of acceptability or the intervention requires bigger adjustments; Red: the majority of intervention participants report the intervention is unacceptable or requires adjustments which cannot be completed.
Completion rate of the outcome measures | Weeks 0 to 10
  The rate of the outcome measures completion will be compared against the following progression criterion to assess the feasibility of outcome measure completion: Green: ≥60%; Amber 40-59%; Red: <40%.
Estimate of between group effect size of the compassion training course intervention compared to control on the primary outcome measure of change in Diabetes Distress Scale scores from baseline (weeks 0-1) to post-intervention (weeks 9 - 10). | Weeks 9 - 10
  The estimated between group effect size of the compassion training intervention compared to control on the primary outcome measure of change in Diabetes Distress Scale scores from baseline (weeks 0-1) to post-intervention (weeks 9-10) will be compared against the following progression criterion to provide a preliminary indicator of effectiveness: Green: effect size in favour of intervention arm and 95% confidence interval for that effect size contains (or is greater than) the minimal clinically important difference (MCID) found in previous research (0.25 or greater). Amber: effect size is in favour of control, but the minimum clinically important difference is included in the 95% confidence interval; Red: effect size is in favour of control, and the minimum clinically important difference is not included in the 95% confidence interval.

SECONDARY OUTCOMES:
Estimate of the between group effect size of compassion training intervention compared to control on change in the Forms of Self-Criticising/ Attacking & Self-Reassuring (FSCRS) Scale from baseline (weeks 0-1) to post-intervention (weeks 9-10). | Weeks 9-10
  The FSCRS is a 22-item self-report measure developed to measure self-criticism and the ability to self-reassure. The scale comprises three subscales: Inadequate-Self, which focuses on feelings of personal inadequacy, Hated-Self, measuring the desire to hurt or punish oneself, and Reassured-Self, which is an ability to reassure and support the self.
Estimate of the between group effect size of compassion training intervention compared to control on change in the External and Internal Shame Scale (EISS) from baseline (weeks 0-1) to post-intervention (weeks 9-10). | Weeks 9-10
  This is an eight-item scale informed by the evolutionary, biopsychosocial model measuring external and internal dimensions of shame. Research shows that individuals with chronic physical health conditions report higher levels of internal and external shame.
Estimate of the between group effect size of compassion training intervention compared to control on change in the Compassionate Engagement and Action Scale (CEAS) from baseline (weeks 0-1) to post-intervention (weeks 9-10). | Weeks 9-10
  The scale has been validated to measure self-compassion through engagement, by assessing engagement with sensitivity, sympathy, non-judgement, empathy, distress tolerance and caring, and self-compassion through action, by balanced reasoning, focusing attention on helpful contexts, actions that alleviate distress and cultivating inner support to alleviate distress. The 13-item sub-scale within the CEAS will be used (compassion to self).

CONTACTS AND LOCATIONS:
Overall Officials: Fergal Jones, PhD, Study Chair — Canterbury Christ Church University; Alan Hebben-Wadey, DClinPsy, Study Director — Canterbury Christ Church University; Jodie Slevin, BSc, Principal Investigator — Canterbury Christ Church University
Locations (2):
- United Kingdom (2):
  - Betsi Cadwaladr University Health Board (BCUHB), Bangor, Wales
  - Barts Health NHS Trust, London

REFERENCES:
- [Background] Banks J, Amspoker AB, Vaughan EM, Woodard L, Naik AD. Ascertainment of Minimal Clinically Important Differences in the Diabetes Distress Scale-17: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Nov 1;6(11):e2342950. doi: 10.1001/jamanetworkopen.2023.42950. PMID 37966840
- See also: Diabetes Distress - Screening Scale (DDS17) — https://healthinnovationnetwork.com/wp-content/uploads/2017/01/Diabetes-Ditress-Screening-Scale.pdf
- See also: The Forms of Self-Criticising/ Attacking & Self-Reassuring Scale (FSCRS) — https://assets-global.website-files.com/641587796769f7a1774bacf4/641587796769f7e8524bb0c6_forms-of-self-criticising-attacking-and-self-reassuring-scale-fscrs.pdf
- See also: Compassionate Engagement and Action Scale (CEAS) — https://cdn.prod.website-files.com/641587796769f7a1774bacf4/641587796769f7da224bb0ec_the-compassionate-engagement-and-action-scales.pdf
- See also: External and Internal Shame Scale (EISS) — https://nationalsocialanxietycenter.com/selfscoring-shame-scale/